CLINICAL TRIAL: NCT01786746
Title: Cognitive Behavioral Therapy (CBT)
Brief Title: Adapting Cognitive Behavioral Therapy (CBT) for Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont McKenna College (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Wei-Chin Hwang, PI, Associate Professor, Claremont McKenna College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH073545 (NIH)
Record Dates: First submitted 2013-02-05; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Major Depression
Keywords: depression; cognitive behavioral therapy; culture; Chinese Americans; psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Psychotherapy (Experimental): Psychotherapy arm that consists of a randomization into 12 session manualized cognitive behavioral therapy or culturally adapted cognitive behavioral therapy for Chinese Americans.
  Interventions: Behavioral: cognitive behavioral therapy; Behavioral: culturally adapted cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy. 12 sessions.
Behavioral: culturally adapted cognitive behavioral therapy — culturally adapted cognitive behavioral therapy for Chinese Americans. 12 sessions.

SUMMARY:
The goals of this study were to a) test whether cognitive behavioral therapy (CBT) is effective in treating depressed Chinese Americans, b) to develop and test the effectiveness of culturally adapt CBT, and c) to test the differential outcomes of the two treatments.

DETAILED DESCRIPTION:
It is now known that ethnic minorities are less likely to receive quality health services and evidence worse treatment outcomes when compared with other groups (IOM, 1999; USDHHS, 2001). Moreover, there continues to be a shortage of systematic investigations examining the efficacy of evidence-based treatments (EBTs) with ethnic minorities, especially among Chinese Americans. Developing interventions that are both empirically grounded and that are culturally sensitive and compatible with Chinese culture is one promising strategy that may improve treatment outcomes for this understudied group. The goal of this study is to culturally adapt a cognitive-behavioral therapy manual for use with depressed Chinese American patients. This study will be among the first to develop a culturally adapted EBT for use with this ethnic group and will involve three study phases. Phase I of the study will focus on modifying and refining a CBT intervention protocol into a manualized treatment for Chinese Americans. Phase two involves a randomized controlled trial (RCT) comparing the effects of the culturally adapted CBT treatment manual with nonadapted CBT. Phase three will involve further refinement of the treatment manual, data analysis, and report writing. Patients will be recruited from an ethnic-specific mental health center that specializes in treating Asian American clientele to participate in the study. Patients will be randomly assigned to either the adapted CBT treatment or the nonadapted CBT treatment. Moreover, feedback from patients and therapists in both conditions will be used to further refine the new treatment manual, provide valuable information about salient issues in treating depressed Chinese Americans, and will provide initial estimates of treatment parameters that will be used in preparing a larger R01 proposal to further test the adapted intervention.

ELIGIBILITY:
Inclusion Criteria:

* depression, Chinese American

Exclusion Criteria:

* bipolar, psychotic disorder, primary substance abuse problem, severe medical conditions that induce depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (Change is being assessed) | baseline, session 4, 8, 12, and three months follow-up
  most commonly used depression rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chin Hwang, PhD, Principal Investigator — Claremont McKenna College
Locations (1):
- Claremont McKenna College, Claremont, California, United States